CLINICAL TRIAL: NCT04795466
Title: Exploratory PLatform Trial on Anti-Inflammatory Agents in Alzheimer's Disease (EXPLAIN-AD): A Randomized, Placebo-controlled, Multicenter Platform Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Various Anti-inflammatory Agents in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease and Mild Alzheimer's Disease
Brief Title: Study of the Efficacy and Safety of Various Anti-inflammatory Agents in Participants With Mild Cognitive Impairment or Mild Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CADPT06A12201
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Alzheimer disease; Mild Cognitive Impairment; Elderly adults; Adults; Memory loss; Dementia; Inflammation; ADPT06
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Memory Disorders; Dementia; Inflammation | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Canakinumab (Experimental): Canakinumab 150 mg SC once every 4 weeks for the first 2 doses followed by 300 mg SC once every 4 weeks for the subsequent 4 doses.
  Interventions: Biological: Canakinumab
- Placebo (Placebo Comparator): Matching placebo sub-cutaneous injections
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Canakinumab — Biological subcutaneous injection
  Other Names: ACZ885
  Arms: Canakinumab
Other: Placebo — Matching placebo subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this platform study was to evaluate the effect of anti-inflammatory agents on cognition in early Alzheimer's disease. Additionally, the safety and tolerability and their effects on central and peripheral inflammation were evaluated. Due to early termination only a single agent could be studied.

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, participant- and investigator-blinded study in participants with either mild cognitive impairment or mild Alzheimer's disease with evidence of peripheral inflammation.

This study was originally planned as a platform study, designed to investigate different agents in a continuous manner. However, due to early termination of the study only one experimental arm was enrolled.

The study included a screening period (Day -60 to Day -8), followed by a baseline period of 7 days (Day -7 to Day -1), a treatment period of 20 weeks (Day 1 to Day 141), a study completion evaluation (EOC1) approximately 30 days after the last agent administration (Day 171) and a second end of cohort visit (EOC2) approximately 140 days after the last agent administration (Day 281).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 45 years and ≤ 90 years at the time of signing the informed consent;
* Participant has a reliable study partner or caregiver can accompany the participant to all visits;
* A diagnosis of probable MCI due to AD or mild AD according to the National Institute on Aging and the Alzheimer's Association (NIA-AA) criteria;
* Confirmed amyloid and tau positivity via CSF sampling performed at screening;
* Mini-Mental State Examination (MMSE) total score of 20 to 24 (inclusive) at screening; OR, MMSE total score of 25-30 (inclusive) plus a DSST score at least 0.5 standard deviation (SD) below normative data at screening.

Exclusion Criteria:

* Use of an investigational agent or an approved product with the intent to modulate inflammation or modulate the course of AD (e.g., Tau ASOs, gene therapy, amyloid or tau vaccine):

  * Previous use of small molecules is allowed if discontinued for at least five half-lives, or at least 30 days from when the expected pharmacodynamic effect has returned to baseline prior to screening, whichever is longer
  * Previous use of monoclonal or polyclonal antibodies or other biologics is allowed if discontinued for at least five half-lives prior to screening
* Current medical or neurological condition that might impact cognition or performance on cognitive assessments, e.g., MCI not due to AD, non-Alzheimer dementia, Huntington's disease, Parkinson's disease, stroke, schizophrenia, bipolar disorder, active major depression, multiple sclerosis (MS), amyotrophic lateral sclerosis (ALS), active seizure disorder, or history of traumatic brain injury associated with loss of consciousness and ongoing residual transient or permanent neurological signs/symptoms including cognitive deficits, and/or associated with skull fracture;
* Diagnosis of vascular dementia prior to screening (e.g., modified Hachinski Ischaemic Scale score > 6 or those who meet the NINDS AIREN criteria for vascular dementia);

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - SUNY at Stony Brook, Stony Brook, New York
- Finland (2):
  - Novartis Investigative Site, Kuopio
  - Novartis Investigative Site, Turku
- Novartis Investigative Site, Reykjavik, Iceland
- United Kingdom (5):
  - Novartis Investigative Site, Plymouth, Devon
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Motherwell
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 sites in 4 different countries
Pre-assignment Details: There was a screening period (Day -60 to Day -8), followed by a baseline period of 7 days (Day -7 to Day -1), before first treatment.
Groups:
- Placebo: Matching placebo subcutaneous injections
Period: Overall Study
Arm/Group | Canakinumab | Placebo
Started | 16 | 18
Pharmacodynamic Analysis Set (The pharmacodynamic (PD) analysis set included all participants with available (total target) PD data and no protocol deviations with relevant impact on (total target) PD data.) | 15 | 18
Completed | 10 | 16
Not Completed | 6 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab | Placebo | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71 (6.53) | 72.4 (6.71) | 71.8 (6.57)
Age, Continuous [Median (Full Range); unit: Years] | 71.5 [58 to 81] | 73.5 [60 to 82] | 72 [58 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 18 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 18 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cognition as Measured by the Neuropsychological Test Battery (NTB) Z-scores
Description: NTB is a composite of multiple neuropsychological tests that provide a thorough assessment of the cognitive domains affected by early Alzheimer's Disease (AD), in particular, memory, executive function, attention and verbal fluency. 5 out of 9 NTB components were administered in the study, Rey Auditory Verbal Learning Test (RAVLT) immediate and delayed scores, Wechsler Memory Scale Digit Span, Controlled Word Association Test (COWAT) and Category Fluency Test (CFT).
  For each component a raw score was converted to z-score that indicates the number of standard deviations away from the mean. Total Z-score was derived by averaging all resulting z-scores. A change from baseline was calculated as post-baseline z-score minus pre-treatment z-score. A zero Z-score means no cognitive change, a negative value indicates decline, and a positive value means improvement.
Time Frame: Baseline and day 171
Population: Participants in the PD analysis set with an available value for the outcome measure. The PD (total target) analysis set for biotherapeutic agents included all participants with available (total target) PD data and no protocol deviations with relevant impact on (total target) PD data.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 16
z-score | 0.225 (0.116) | 0.156 (0.0905)
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; NTB Total z-score - day 171; Test type: Superiority; p = 0.6386, Mixed Models Analysis; Least square mean difference = 0.069, 90% CI 2-sided [-0.178 to 0.316], Standard Error of Mean 0.1442

2. Secondary Outcome: Change From Baseline in Memory as Measured by the Total Composite NTB Memory Z-score
Description: Total Neuropsychological Test Battery memory composite score is a "memory function" score composed of the NTB RAVLT immediate and delayed scores.
  For each component a raw score was converted to z-score that indicates the number of standard deviations away from the mean. Total Z-score was derived by averaging the two resulting z-scores. A change from baseline was calculated as post-baseline z-score minus pre-treatment z-score. A zero Z-score means no cognitive change, a negative value indicates decline, and a positive value means improvement.
Time Frame: Baseline and day 171
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score change from baseline
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 16
z-score change from baseline | 0.461 (0.1382) | 0.463 (0.1062)
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Memory function - day 171; Test type: Superiority; p = 0.9917, Mixed Models Analysis; Least squares mean difference = -0.002, 90% CI 2-sided [-0.300 to 0.296], Standard Error of Mean 0.1739

3. Secondary Outcome: Change From Baseline in Executive Function as Measured by the Total Composite NTB Executive Function Z-score
Description: The total Neuropsychological Test Battery executive function composite score is an "executive function" score composed of the NTB Wechsler Memory Scale Digit Span, COWAT, and CFT.
  For each component a raw score was converted to z-score that indicates the number of standard deviations away from the mean. Total Z-score was derived by averaging the two resulting z-scores. A change from baseline was calculated as post-baseline z-score minus pre-treatment z-score. A zero Z-score means no cognitive change, a negative value indicates decline, and a positive value means improvement.
Time Frame: Baseline and day 171
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score change from baseline
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 16
z-score change from baseline | 0.111 (0.1492) | -0.075 (0.1251)
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Executive function- day 171; Test type: Superiority; p = 0.3510, Mixed Models Analysis; least squares mean difference = 0.186, 90% CI 2-sided [-0.148 to 0.520], Standard Error of Mean 0.1958

4. Secondary Outcome: Change From Baseline in Digit Symbol Substitution Test (DSST) Score - CANTAB
Description: The DSST is an attention-demanding component of the Wechsler Adult Intelligence Scale-IV.
  The DSST score is the number of digits coded correctly in a fixed amount of time. The DSST has a minimum of "0" correct responses and does not have a maximum; a higher number on the DSST represents better performance
  The test was administered using CANTAB web based testing
Time Frame: Baseline and day 171
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: DSST score change from baseline
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 16
DSST score change from baseline | 1.96 (1.37) | 2.45 (1.13)
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; DSST - day 171; Test type: Superiority; p = 0.7870, Mixed Models Analysis; Repeated measures analysis = -0.49, 90% CI 2-sided [-3.56 to 2.58], Standard Error of Mean 1.80

5. Secondary Outcome: Change From Baseline in Neuropsychiatric Symptoms as Measured by the Neuropsychiatric Inventory (NPI) Total Score
Description: Neuropsychiatric Inventory (NPI) total score is globally recognized and the most frequently used assessment of neuropsychiatric symptoms in AD trials. NPI covers twelve neuropsychiatric domains. For each domain there are four scores, frequency (rated 1-4), severity (rated 1-3), domain total score (frequency x severity) and caregiver distress score (rated 0-5).
  The NPI total score was calculated by adding 12 domain total scores together, and ranges from 0 to 144, with higher values indicating greater severity.
Time Frame: Baseline and day 171
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: NPI total score change from Baseline
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 16
NPI total score change from Baseline | -1.4 (7.76) | 2.9 (8.68)

6. Secondary Outcome: Change From Baseline in Neuropsychiatric Symptoms Associated Distress as Measured by the Neuropsychiatric Inventory Caregiver Distress (NPI-D) Score
Description: Neuropsychiatric Inventory (NPI) total score is globally recognized and the most frequently used assessment of neuropsychiatric symptoms in AD trials. NPI covers twelve neuropsychiatric domains. For each domain there are four scores, frequency (rated 1-4), severity (rated 1-3), domain total score (frequency x severity) and caregiver distress score (rated 0-5).
  The caregiver distress score (NPI-D) was calculated by adding together the scores of the 12 individual NPI distress questions, and ranges from 0 to 60, with higher values indicating greater severity.
Time Frame: Baseline and day 171
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: NPI-D score change from Baseline
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 16
NPI-D score change from Baseline | -2.7 (7.70) | 1.2 (5.74)

7. Secondary Outcome: Change From Baseline in Mean eNeuropsychiatric at Home Caregiver Assessment Score
Description: Neuropsychiatric Inventory (NPI) total score is globally recognized and the most frequently used assessment of neuropsychiatric symptoms in AD trials. NPI covers twelve neuropsychiatric domains. For each domain there are four scores, frequency (rated 1-4), severity (rated 1-3), domain total score (frequency x severity) and caregiver distress score (rated 0-5).
  The eNeuropsychiatric at-home assessment was calculated the same way as the in-clinic NPI by adding the12 domain total scores together. The eNeuropsychiatric at-home assessments were completed more frequently than the single time-point in-clinic NPI assessment and the scores averaged. It ranges from 0 to 144, with higher values indicating greater severity.
Time Frame: Baseline, day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 12
scores on a scale | 0.983 (3.7904) | -1.094 (1.7083)

8. Secondary Outcome: Change From Baseline in Everyday Cognition Scale (ECog) Total Score
Description: Everyday Cognition (ECog) scale measures cognitively-relevant everyday abilities and is comprised of 39 items covering six cognitively-relevant domains: Everyday Memory, Everyday Language, Everyday Visuospatial Abilities, Everyday Planning, Everyday Organization, and Everyday Divided Attention. Each item is scored on a 4 point scale (1=better or no change compared to 10 years earlier, 2=questionable/occasionally worse, 3=consistently a little worse, 4=consistently much worse). An "I don't know" response is also included, in that case the item is not included in the calculation.
  The total ECog score is calculated as the sum of all 39 items, and ranges from 0 to 156. Lower total ECog scores indicate better performance.
Time Frame: Baseline and day 171
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ECog total score change from Baseline
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 10 | 16
ECog total score change from Baseline | 1.2 (14.26) | 3.4 (11.79)

9. Secondary Outcome: Change From Baseline in eCognitive Testing Scores - SWM Between Errors
Description: Spatial Working Memory (SWM) is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. A trial begins with several colored squares (boxes) being shown on the screen. The overall aim is that the subject should find a blue 'token' in each of the boxes and use them to fill up an empty column. The subject must touch each box in turn until one opens with a blue 'token' inside (a search). Returning to an empty box already sampled on this search is an error.
  SWM between errors is the number of times the subject incorrectly revisits a box in which a token has previously been found. It starts at 0 without a maximum limit with higher scores indicating a worse outcome.
Time Frame: Baseline, day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SWMBE score change from baseline
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 9 | 12
SWMBE score change from baseline | -1.56 (6.018) | -1.83 (4.910)

10. Secondary Outcome: Change From Baseline in eCognitive Testing Scores - SWM Strategy
Description: Spatial Working Memory (SWM) is a test of the subject's ability to retain spatial information and to manipulate remembered items in working memory. A trial begins with several colored squares (boxes) being shown on the screen. The overall aim is that the subject should find a blue 'token' in each of the boxes and use them to fill up an empty column. The subject must touch each box in turn until one opens with a blue 'token' inside (a search). Returning to an empty box already sampled on this search is an error.
  SWM Strategy is the number of times a subject begins a new search pattern from the same box they started with previously. If they always begin a search from the same starting point, we infer that the subject is employing a planned strategy for finding the tokens. SMW strategy ranges from 3 to 26, a low score indicates high strategy use, they always begin the search from the same box, and a high score indicates that they are beginning their searches from many different boxes.
Time Frame: Baseline, day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 9 | 12
scores on a scale | -0.28 (1.149) | -0.92 (1.459)

11. Secondary Outcome: Change From Baseline in eCognitive Testing Scores - MTS Proportional Slowing 8-2 Patterns
Description: Match to Sample Visual Search (MTS) assesses attention and visual searching, with a speed accuracy trade-off. The participant is shown a complex visual pattern in the middle of the screen. After a brief delay, a varying number of similar patterns are shown in a circle of boxes around the edge of the screen. Only one of these patterns matches the pattern in the center of the screen, and the participant must indicate which it is by selecting it.
  MTS proportional slowing 8-2 patterns is the difference in mean time between presentation of the response stimulus options and the subject selecting the correct box on their first attempt on the 8 pattern assessment trials compared to the 2 pattern assessment trials. It starts at 0 without a maximum limit, and with higher scores indicating a worse outcome.
Time Frame: Baseline, day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change from baseline in milliseconds
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 9 | 12
Change from baseline in milliseconds | 143.780 (2871.0641) | 77.573 (2824.3325)

12. Secondary Outcome: Change From Baseline in eCognitive Testing Scores - PAL First Attempt Memory Score
Description: Pair associated learning (PAL): tests participants' visual memory/new learning using patterns randomly displayed in boxes on a screen. Participants are to touch the box where patterns first appeared.
  PAL first attempt memory score is the number of times a subject choses the correct box on their first attempt when recalling the pattern locations. Ranges from 0 to 20 with higher score indicates a better outcome.
Time Frame: Baseline, day 85
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PAL score change from baseline
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 9 | 12
PAL score change from baseline | -0.17 (2.716) | 0.08 (3.059)

13. Secondary Outcome: Change From Baseline in Microglia Activation as Measured by Positron-Emission Tomography-Translocator Protein 18kDa - Microglia Activation
Description: Positron-Emission Tomography-Translocator Protein 18kDa-microglia activation (PET TSPO) is considered a marker of central inflammation (a marker for activated microglia and astrocytes) and the signal strength has been shown to correlate with worsening clinical severity in participants with MCI or AD, measures of cognition and various clinical scores. Relative % change from baseline in volume of distribution (Vt) of the radio tracer for TSPO after treatment.
  Since only one participant completed day 85 PET TSPO, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: Baseline and day 85
Population: Participants in the PD analysis set with an available value for the outcome measure. The PD (total target) analysis set for biotherapeutic agents included all participants with available (total target) PD data and no protocol deviations with relevant impact on (total target) PD data.
  PET TSPO inferential analysis could only be performed if the number of participants with data allowed the analysis without compromising patient privacy/confidentiality.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 0 | 1
Percent change from baseline |  | NA (NA) — Only one participant completed day 85 PET TSPO, Data not reported in order to protect and maintain participant privacy/confidentiality.

14. Secondary Outcome: Serum Pharmacokinetic Concentrations of Canakinumab
Description: Serum pharmacokinetic pre-dose concentrations of CanakinumabConcentrations below the LLOQ were reported as "zero".
Time Frame: Baseline, day29, day 57, day 85, day 141, day 171
Population: Participants in the pharmacokinetic (PK) analysis set who received Canakinumab. The PK analysis set included all participants with at least one available valid (i.e., not flagged for exclusion) PK concentration measurement, who received any study drug and with no protocol deviations that impact PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Canakinumab
Number analyzed (Participants) | 16
ng/mL
  Baseline: number analyzed (Participants) | 14
  Baseline | 0.0 (0.00)
  Day 29 | 8921.3 (2721.47)
  Day 57: number analyzed (Participants) | 13
  Day 57 | 14230.8 (4712.07)
  Day 85: number analyzed (Participants) | 12
  Day 85 | 26575.0 (10216.93)
  Day 141: number analyzed (Participants) | 11
  Day 141 | 34000.0 (11288.67)
  Day 171: number analyzed (Participants) | 10
  Day 171 | 33170.0 (6825.45)

15. Secondary Outcome: Total Target (IL-1 Beta) Concentration in Serum and CSF
Description: Serum and CSF samples were obtained and evaluated for total target concentrations (the sum of free and drug-bound target) as a pharmacodynamic (PD) marker for target engagement.
Time Frame: Baseline, day 29, day 57, day 85, day 141, day 171 for serum concentrations and Baseline and day 85 for CSF concentrations
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 15 | 18
pg/mL
  Serum - Baseline: number analyzed (Participants) | 13 | 18
  Serum - Baseline | 0.000 (0.0000) | 0.000 (0.0000)
  Serum - Day 29 | 12.632 (4.4949) | 0.000 (0.0000)
  Serum - Day 57: number analyzed (Participants) | 13 | 17
  Serum - Day 57 | 20.818 (10.2918) | 0.000 (0.0000)
  Serum - Day 85: number analyzed (Participants) | 11 | 16
  Serum - Day 85 | 23.291 (5.2984) | 0.000 (0.0000)
  Serum - Day 141: number analyzed (Participants) | 11 | 16
  Serum - Day 141 | 44.473 (58.3963) | 0.000 (0.0000)
  Serum - Day 171: number analyzed (Participants) | 10 | 16
  Serum - Day 171 | 28.460 (18.4483) | 0.000 (0.0000)
  CSF - Baseline | 0.000 (0.0000) | 0.000 (0.0000)
  CSF - Day 85: number analyzed (Participants) | 12 | 15
  CSF - Day 85 | 0.000 (0.0000) | 0.023 (0.0883)

16. Secondary Outcome: Number of Participants With Anti-agent Antibodies in Serum
Description: Number of participants with anti-agent antibodies in serum. Immunogenicity (IG) was assessed in serum of all participants treated with biotherapeutic drug.
Time Frame: Baseline, day 85, day 171
Population: Participants in the safety analysis (SA) set who received Canakinumab. The SA set included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 16
Participants
  Baseline: POSITIVE | 0
  Baseline: NEGATIVE | 16
  Day 85: number analyzed (Participants) | 12
  Day 85: POSITIVE | 0
  Day 85: NEGATIVE | 12
  Day 171: number analyzed (Participants) | 10
  Day 171: POSITIVE | 0
  Day 171: NEGATIVE | 10

17. Secondary Outcome: Number of Participants Who Experience Adverse Events and Serious Adverse Events
Description: Clinically significant abnormalities of laboratory values, physical findings, electrocardiogram findings and other safety assessments were recorded as adverse events if the findings meet the defined criteria for adverse events.
  AE grades to characterize the severity of the AEs were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5. For CTCAE, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE
Time Frame: From first dose up to approximately 140 days post last dose (day 281)
Population: The safety analysis set included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 16 | 18
Participants
  Participants with at least one AE | 14 | 16
  Participants with grade 1 AEs | 14 | 16
  Participants with grade 2 AEs | 6 | 6
  Participants with grade 3 AEs | 1 | 0
  Participants with study drug related AEs | 4 | 5
  Participants with serious AEs | 2 | 1
  Participants with AEs leading to treatment discontinuation | 3 | 1
  Participants with study drug related AEs leading to treatment discontinuation | 1 | 0

ADVERSE EVENTS:
Time Frame: From first dose up to approximately 140 days post last dose (day 281)
Groups:
- Total: Total
Arm/Group | Canakinumab | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18 | 0/34
Serious Adverse Events (participants affected / at risk) | 2/16 | 1/18 | 3/34
Other Adverse Events (participants affected / at risk) | 13/16 | 16/18 | 29/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=16) | Placebo (N=18) | Total (N=34)
COVID-19 (Infections and infestations) | 1 | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab (N=16) | Placebo (N=18) | Total (N=34)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Sensitisation (Immune system disorders) | 0 | 1 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Otitis externa (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 3
Vaginal infection (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Immunisation reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 2 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Lipase increased (Investigations) | 1 | 2 | 3
Weight decreased (Investigations) | 1 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 2
Headache (Nervous system disorders) | 0 | 1 | 1
Intention tremor (Nervous system disorders) | 0 | 1 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 2
Irritability (Psychiatric disorders) | 1 | 0 | 1
Persecutory delusion (Psychiatric disorders) | 1 | 0 | 1
Procedural anxiety (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 4 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT04795466/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT04795466/SAP_001.pdf